CLINICAL TRIAL: NCT04890327
Title: Clinical Utility of a Web-based Tool for Collection of Family Health History and Risk-assessment in Patients Presenting to a Gynecologic Oncology Clinic
Brief Title: Web-based Family History Tool
Acronym: Progeny
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1612017795
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Gynecologic Cancer; Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Patient presents to new Gynecologic Oncology appointment, family health history is collected by the physician during the clinic visit. Both the subject and physician complete assessment survey at the completion of clinic visit. Subject's medical record reviewed 6 months following study enrollment to determine subject's diagnosis, whether or not subject underwent genetic counseling and/or genetic testing and review genetic testing results.
- Office (Experimental): Patient presents to new Gynecologic Oncology appointment, subject is given access to a desk top computer in office and instructed to complete web-based family health history tool. Physician reviews results of patients web-based family health history tool.Subject and physician complete assessment survey at the completion of clinic visit. Subject's medical record reviewed 6 months following study enrollment to determine subject's diagnosis, whether or not subject underwent genetic counseling and/or genetic testing and review genetic testing results.
  Interventions: Other: Web-based family health history tool
- Home (Experimental): Patient is emailed a link containing web-based family health history tool prior to presenting for new Gynecologic Oncology appointment. Physician reviews results of patients web-based family health history tool. Subject and physician complete assessment survey at the completion of clinic visit. Subject's medical record reviewed 6 months following study enrollment to determine subject's diagnosis, whether or not subject underwent genetic counseling and/or genetic testing and review genetic testing results.
  Interventions: Other: Web-based family health history tool

INTERVENTIONS:
Other: Web-based family health history tool — Web-based tool that collects subject's family health history through a series of questions and generates a pedigree which documents a risk assessment report for the physician to use. The risk assessment report uses standard, validated risk scores including GAIL , CLAUS, BRCAPRO which measure breast cancer risk, and MMRPRO which measures endometrial cancer risk, MELAPRO which measures melanoma cancer risk, and PANCPRO which measures pancreatic cancer risk
  Arms: Home; Office

SUMMARY:
The purpose of this pilot study is to determine if a web-based tool that collects family health history is useful for patients being seen in a gynecologic oncology office setting. This research study is being done because collecting a comprehensive family health history is critical as it allows physicians to appropriately refer patients for genetic counseling and genetic testing. However, prior research indicates that the family health history collected in clinical settings is often inadequate to truly assess the risk of genetic disease. Therefore we plan to explore a web-based program that guides patients through the collection of their family health history and uses this information to create clear concise pedigrees (family tree information) and risk assessment models that can be used by a physician during the office visit.

DETAILED DESCRIPTION:
Patients presenting for a new patient visit with a gynecologic oncologist will be randomized to one of three methods of collection of family health history (Arm 1 - standard of care consisting of interview with the physician; Arm 2 - completion of a web-based family health history tool completed in the clinic waiting room on a computer; Arm 3 - completion of a web-based family health history tool completed prior to the visit and accessed by an email link). A new 4th arm was added with 200 chart reviews to retrospectively look back at how previous family health history was taken for new patients in 2019. The study will evaluate the quality of the family health history collected, the resulting referral to genetic services and patient and physician satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Female > 18 years of age. Scheduled for new patient visit with one of the gynecologic oncologists at Weill Cornell Medicine (Melissa Frey MD, Kevin Holcomb MD, Evelyn Cantillo MD, Eloise Chapman MD).

Exclusion Criteria:

Subjects who cannot communicate in English as the FHH collection tool and surveys are available only in English.

Subjects who were adopted and have no information about their family health history.

Subjects who do not present for the new patient visit.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with high quality family health history (FHH) | Anytime between 18 - 24 months
  To compare the amount of subjects with a high quality family health history in each of the study arms that properly assesses disease risk. Currently FHH in a gynecologic oncology clinic setting is inadequate to assess disease risk. The use of a web-based FHH collection tool that also offers the providers with a risk assessment tool may address these challenges and increase the comprehensiveness of FHH collection and risk assessment in the gynecologic oncology clinic.
  For a pedigree to be considered high quality, at least one individual in the pedigree must meet all quality criteria ("high quality relative").
  1. Three generations of relatives
  2. Relatives' lineage (e.g. paternal or maternal side)
  3. Relatives' gender
  4. An up-to-date FHH
  5. Pertinent negatives in FHH noted (i.e. no FHH of cancer)
  6. Age of disease onset in affected relatives
  7. For deceased relatives - the age of death
  8. For deceased relatives - the cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Frey, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No